CLINICAL TRIAL: NCT06082635
Title: A Multi-centered, Randomized, Open-label Phase III Study to Evaluate the Efficacy and Safety of TGRX-326 Comparing With Crizotinib in Patients of Advanced ALK-positive or Metastatic Non-Small Cell Lung Cancer
Brief Title: TGRX-326 Chinese Phase III for Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-326-3001-NSCLC-CN
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TGRX-326 (Experimental): Subjects to be treated with the investigational drug TGRX-326 at 60 mg once day in 28-day cycles.
  Interventions: Drug: TGRX-326
- Crizotinib (Active Comparator): Subjects to be treated with the active control drug crizotinib at 250 mg twice day in 28-day cycles.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: TGRX-326 — Subjects will be treated with the investigational drug TGRX-326 at 60 mg once a day in 28-day cycles
  Other Names: TGRX-326 QD (once a day)
  Arms: TGRX-326
Drug: Crizotinib — Subjects will be treated with the control drug crizotinib at 250 mg twice a day in 28-day cycles
  Other Names: Crizotinib 250 mg BID (twice a day)
  Arms: Crizotinib

SUMMARY:
This is a multi-center, randomized, open-label, Phase III clinical trial which compares the safety and efficacy of TGRX-326 with crizotinib in patients with ALK-positive advanced or metastatic NSCLC

DETAILED DESCRIPTION:
This Phase III study aims to evaluate the safety profile and efficacy profile in patients with ALK-positive advanced or metastatic NSCLC and to compare the efficacy and safety of TGRX-326 with that of crizotinib. The primary purpose of this study is to evaluate and compare the efficacy profile of TGRX-326 with crizotinib, with progression-free survival (PFS) as evaluated by independent review committee (IRC) as end point. Secondary objectives include comparing efficacy profile of other endpoints and safety profiles of the investigational drug with crizotinib. Exploratory objective includes the evaluation of population pharmacokinetic (PK) profile of TGRX-326 and efficacy of TGRX-326 in ALK-positive advanced NSCLC patients determined as progressive disease after crizotinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing to follow the treatment protocol and visit schedule, and participate in the study with the ICF signed;
* ≥ 18 years of age on the day of ICF signing, regardless of gender.
* Diagnosed as incurable stage IIIB - IV ALK-positive NSCLC;
* Providing prior ALK positive test results at screening;
* Naïve to ALK-inhibitor; patients could be intolerant or have progressive disease from previous first-line chemotherapy;
* Patients could have metastases to central nervous system at screening if the condition is asymptomatic, stable or completely recovered;
* At least one measurable lesion;
* An ECOG PS score within 0-2;
* Adequate bone marrow, liver, kidney, coagulation and pancreatic functions;
* Expected survival ≥ 3 months;
* Willing to take effective contraceptive measures (for men of reproductive potential and women of reproductive age only) from ICF signing to 6 months after last administration of the investigational drug. Women of reproductive age include women before menopause and within 1 year after menopause; those women must have a negative pregnancy test ≤ 7 days prior to the first dose of the investigational drug.

Exclusion Criteria:

* Known hypersensitivity to any of the active ingredients or excipients of TGRX-326 or crizotinib pills; or a history of severe allergic reactions;
* Having another type of cancer except for lung cancer;
* Radiotherapy within 14 days prior to the first dose;
* Received other systemic anti-tumor treatment within 4 weeks prior to the first dose, or is within 5 half-lives of the said treatment; received traditional Chinese medicine indicated for anti-tumor purposes within 14 days prior to the first dose;
* Major surgery within 4 weeks prior to the first dose;
* Spinal cord compression caused by tumor, unless the subject achieves significant pain control and full recovery of neurological function within 4 weeks prior to the first dose.
* Abnormal gastrointestinal function that affect absorption within the past 6 months;
* History of active pneumonia or clinically significant interstitial pneumonia, or radiation or drug-induced lung disorder with treatment needs;
* Cardiac insufficiency;
* Abnormal and clinically significant QTc on ECG or need of concomitant use of any drug known to prolong QT interval and cause torsades de pointes;
* Uncontrolled hypertension after drug treatment;
* Uncontrolled hyperglycaemia, acute attack of cholelithiasis, and susceptibility to acute pancreatitis;
* Severe or uncontrolled systemic diseases causing expected intolerance to the investigational drug as judged by the investigator;
* Toxic reactions associated with prior surgery and prior antineoplastic therapies that have not recovered and may affect the subject safety as assessed by the investigator.
* Clinically significant active bacterial, fungal or viral infections, including a positive result for hepatitis B surface antigen and HBV DNA ≥ ULN, one or more positive results for hepatitis C antibody or HIV antibody, or the presence of any uncontrolled infection.
* Use of strong CYP3A4 inducers or inhibitors or CYP3A4 substrates with a narrow therapeutic window within two weeks prior to the first dose of the investigational drug;
* Pregnant and breastfeeding female;
* Women of childbearing age who are unwilling or unable to use acceptable methods for contraception during the entire treatment period in the trial and within 6 months after the last dose of the investigational drug (women of childbearing age include: any one with menarche, and those who have not received successful artificial sterilization [hysterectomy, bilateral fallopian tube ligation, or bilateral oophorectomy] or premenopausal women); a fertile male patient who is unwilling or unable to take effective contraceptive measures, and whose partner is a woman of childbearing age;
* Being involved in other clinical studies (except for the non-interventional phase of interventional clinical study, such as survival follow-up period); less than 4 weeks from the end of the dose of other investigational drug to the first dose of the investigational drug or 5 half-lives of the previous drug, whichever is shorter;
* Any mental or cognitive disorders which may limit subjects' understanding and implementation of the informed consent form;
* Other situations, such as poor compliance, which are considered by the investigator to be not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by independent review committee (IRC) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  PFS defined by the time from randomization to progressive disease or death of any cause; PFS as evaluated by independent review committee (IRC).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by investigator | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  PFS defined by the time from randomization to progressive disease or death of any cause; PFS as evaluated by investigator.
One-year Progression Free Survival (PFS) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  One-year PFS defined by the time from randomization to progressive disease or death of any cause, with data collection up to 1 year from randomization; one-year PFS as evaluated by investigator or IRC.
Objective Response Rate (ORR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  ORR defined by the ratio of patients who reached the treatment response; ORR as evaluated by independent review committee (IRC) and investigator
Duration of Response (DOR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  DOR defined as the duration from first occurence of treatment response to progressive disease/relapse; DOR as evaluated by IRC and investigator
Disease Control Rate (DCR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  DCR defined by the ratio of patients who reached the treatment response or maintained as stable disease; DCR as evaluated by IRC and investigator
Time to Response (TTR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  TTR defined by the time from the start of treatment to the first ORR; TTR as evaluated by IRC and investigator
Intracranial Objective Response Rate (IC-ORR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  IC-ORR defined by the ratio of patients who reached the intracranial treatment response; ORR as evaluated by IRC and investigator.
Intracranial Disease Control Rate (IC-DCR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  IC-DCR defined by the ratio of patients who reached the treatment response intracranially or maintained as stable disease; IC-DCR as evaluated by IRC and investigator
Intracranial Duration of Response (IC-DOR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  IC-DOR defined as the duration from first occurrence of Intracranial treatment response to progressive disease/relapse; DOR as evaluated by IRC and investigator
Intracranial Time to Response (IC-TTR) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  IC-TTR defined by the time from the start of treatment to the first IC-ORR; TTR as evaluated by IRC and investigator
Intracranial Progression Free Survival (IC-PFS) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  IC-PFS defined by the time from randomization to progressive disease or death of any cause in patients with intracranial lesions; PFS as evaluated by IRC and investigator.
Overall Survival (OS) | Every 8 weeks between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 28 days); an average of 1.5 years
  OS defined by the time from randomization to death of any cause
Adverse Events (AEs) | At Screening; Day 1 of every Cycle (each cycle is 28 days) until end of study
  To record and analyze subjects with adverse events (AEs)
Serious Adverse Events (SAEs) | At Screening; Day 1 of every Cycle (each cycle is 28 days) until end of study
  To record and analyze subjects with serious adverse events (SAEs)

OTHER OUTCOMES:
Plasma Cmax | Day 1 of Cycle 2, 3 and 5 (each cycle is 28 days)
  To measure plasma TGRX-326 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No